CLINICAL TRIAL: NCT03014180
Title: Clinical Evaluation of LEft VEntricular Auto Threshold Algorithm
Brief Title: Clinical Evaluation of LEft VEntricular Auto Threshold Algorithm (LEVEA)
Acronym: LEVEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LivaNova (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPTL01
Record Dates: First submitted 2016-10-11; First posted 2017-01-09 (Estimated); Results first posted 2019-05-28 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2018-09

CONDITIONS: Heart Failure
Keywords: Heart failure, CRT
MeSH Terms: conditions — Heart Failure; Creatine deficiency, X-linked

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- "In-Clinic LVAT" (Experimental): All subject prior to study enrollment has been implanted with a CRT-D device. During follow-ups, under the supervision of the physician, the algorithm embeded in the device is activated with a password. The feature is deactivated at the end of each follow-up.
  Interventions: Device: "In-Clinic LVAT"

INTERVENTIONS:
Device: "In-Clinic LVAT" — Algorithm offers automatic threshold measurement of differents vectors of left ventricular stimulation.
  Other Names: Activation of an algorithm in CRT-D device

SUMMARY:
The purpose of the LEVEA study is to assess the performances of a new automatic left ventricular auto threshold (LVAT) algorithm (In-Clinic LVAT algorithm) when used by physicians during in-hospital follow-up.

DETAILED DESCRIPTION:
"In-Clinic LVAT" feature is a non CE-marked feature designed to be activated by the physician during 2 hospital follow-ups:

* first visit: planned to be conducted 15 days maximum after inclusion
* second visit: planned to be conducted between 1 and 3 months after the first visit The evaluation consists in the comparison between the threshold value provided by the algorithm and the threshold value obtained manually by the physician.

ELIGIBILITY:
Inclusion Criteria:

* Subject already implanted (de-novo, upgrade or replacement) according to the relevant ESC Guidelines [1]:

  * With IS1 Platinium SonR CRT-D (models 1811, 1841, CE-marked) for maximum of 5 days or;
  * With IS4 Platinium SonR CRT-D (model 1844, CE-marked).
* Right atrial, right and left ventricular leads must be implanted. Only bipolar and quadripolar for Left Ventricular lead.
* Reviewed, signed and dated informed consent.

Exclusion Criteria:

* Subject included in another clinical study that could confound the results of this study;
* Malfunction or dislodgment of right atrial, right and left ventricular implanted leads;
* Subject diagnosed with permanent atrial fibrillation;
* Known pregnancy;
* Minor age;
* Under protection or guardianship;
* Unavailability for scheduled follow-up or refusal to cooperate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2017-08-17 (Actual); Study Completion 2017-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Mansourati, Pr, Principal Investigator — CHRU de Brest, FRANCE.
Locations (1):
- CHRU Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects have been included from Feb 16, 2017 to June 2, 2017.
Pre-assignment Details: All the 60 patients were assigned to the treatment arm.
Groups:
- "In-Clinic LVAT": 60 patients were included in the single-arm study. The Left Ventricular auto threshold (LVAT) algorithm test was performed at the 2 study visits M0 and M1.
Period: Overall Study
Arm/Group | "In-Clinic LVAT"
Started | 60
Completed | 58
Not Completed | 2
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Groups:
- "In-Clinic LVAT": Single-arm study design: all the 60 patients were assigned to the treatment arm.
Arm/Group | "In-Clinic LVAT"
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (8.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 60
Region of Enrollment [Number; unit: participants]
  France | 43
  Spain | 9
  Germany | 8
Type of device implanted [Count of Participants; unit: Participants]
  IS1 | 24
  IS4 | 36

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Successful"In-Clinic LVAT" Test
Description: The success rate is defined as the equivalence between the value measured by the algorithm and the measure obtained manually by the physician on 5 identified pacing vectors during the visit among at least 231 LV tests.
Time Frame: 0-3 months post inclusion
Population: Complete LV vector test: test was performed (not aborted or interrupted) and a threshold value is provided by the algorithm.
  Successful LV Vector Test: LV threshold value provided by the algorithm compared to the manual threshold is considered "Successful" if the difference is within ± 2 step
Measure: Number (95% Confidence Interval); unit: percentage of successful LVAT test
Units Other Than Participants: Completed LV vector tests
Groups:
- In-clinic LVAT: Patients assigned to the single-arm treatment LVAT. LVAT test performed at M0 and M1 visits.
Arm/Group | In-clinic LVAT
Number analyzed (Participants) | 56
Number analyzed (Completed LV vector tests) | 262
percentage of successful LVAT test | 94.66 [90.66 to 97.31]

2. Secondary Outcome: Percentage of Accurate "In-Clinic LVAT" Test Assessed by an Independent Reviewer
Description: This endpoint is the number of accurate determination of the pacing threshold value provided by the algorithm feature and an independent reviewer, on all available LV pacing vectors at first visit.
  An independent reviewer assessed all LV pacing threshold values provided by the algorithm at M0 visit and in all tested configurations
Time Frame: 0-15 days post inclusion
Population: Completed LV Vector Test: test was performed (not aborted or interrupted) and a threshold value is provided by the algorithm.
  Accurate LV Vector Test: The LV threshold value provided by the algorithm compared to the reviewer assessment is considered accurate if the difference is within ± 1 step.
Measure: Number (95% Confidence Interval); unit: Percentage of accurate determination
Units Other Than Participants: Number of completed LV Vector Tests
Groups:
- In-clinic LVAT: Patients assigned to the single-arm treatment LVAT. LVAT test performed at M0 visit.
Arm/Group | In-clinic LVAT
Number analyzed (Participants) | 55
Number analyzed (Number of completed LV Vector Tests) | 1301
Percentage of accurate determination | 99.31 [98.59 to 99.72]

3. Secondary Outcome: Percentage of Successful of "In-Clinic LVAT" Test at M0 Visit
Description: The success rate of "In-Clinic LVAT" feature for all available LV pacing vectors at first follow-up (M0 visit). The method of analysis is similar to the primary endpoint.
Time Frame: 0-15 days post inclusion
Population: Completed LV vector Test: test was performed (not aborted or interrupted) and a threshold value is provided by the algorithm.
  Successful LV Vector Test: LV threshold value provided by the algorithm compared to the manual threshold is considered "Successful" if the difference is within ± 2 steps
Measure: Number (95% Confidence Interval); unit: Percentage of successful LVAT test
Units Other Than Participants: Number of completed LV Vector Tests
Groups:
- In-clinic LVAT: Patients assigned to the single-arm treatment LVAT at M0 visit.
Arm/Group | In-clinic LVAT
Number analyzed (Participants) | 55
Number analyzed (Number of completed LV Vector Tests) | 1193
Percentage of successful LVAT test | 90.86 [88.82 to 92.65]

4. Secondary Outcome: Percentage of Successful "In-Clinic LVAT" Test at M1 Visit
Description: The success rate of "In-Clinic LVAT" feature for all available LV pacing vectors at second follow-up . The method of analysis is similar to the primary endpoint
Time Frame: 1-3 months after first visit
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Pecentage of successful LVAT test
Units Other Than Participants: Number of completed LV Vector Tests
Groups:
- In-clinic LVAT: Patients assigned to the single-arm treatment LVAT at M1 visit.
Arm/Group | In-clinic LVAT
Number analyzed (Participants) | 56
Number analyzed (Number of completed LV Vector Tests) | 1217
Pecentage of successful LVAT test | 92.03 [90.12 to 93.68]

5. Secondary Outcome: Percentage of Eligible Subjects to LVAT Feature
Description: Identification of the number of subjects who were "eligible" to receive the feature at M0 or M1 visit
Time Frame: 0-3 months post inclusion
Population: Eligible subjects: Number of subjects with at least one complete LV Vector Test at M0 or M1 visits
Measure: Number; unit: Percentage of eligible subjects
Arm/Group | In-clinic LVAT
Number analyzed (Participants) | 57
Percentage of eligible subjects | 98.25

6. Secondary Outcome: Safety of the LVAT Algorithm
Description: Reporting of SAEs, device deficiencies and any suspect behaviour of the algorithm.
Time Frame: 0-3 months post inclusion
Population: Included population
Measure: Number; unit: Event
Groups:
- Secondary Endpoint: All serious adverse events and device deficiency during in-clinic LVAT test.
Arm/Group | Secondary Endpoint
Number analyzed (Participants) | 60
Event | 6

ADVERSE EVENTS:
Time Frame: 0-3 months post inclusion
Description: SAE and device deficiency were collected through the study duration and AE was collected at each study visit.
Groups:
- In-Clinic LVAT: All serious adverse events and device deficiency during in-clinic LVAT test.
Arm/Group | In-Clinic LVAT
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 6/60
Other Adverse Events (participants affected / at risk) | 0/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | In-Clinic LVAT (N=60)
Cardiac decompensation (Cardiac disorders) | 2 (2)
Heart failure worsening (Cardiac disorders) | 1 (1)
Bleeding (Injury, poisoning and procedural complications) | 2 (2)
Embolization (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2016-09-29): https://cdn.clinicaltrials.gov/large-docs/80/NCT03014180/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-20): https://cdn.clinicaltrials.gov/large-docs/80/NCT03014180/SAP_001.pdf